CLINICAL TRIAL: NCT01898325
Title: Assessment Of Liver and Spleen Fibrosis in Patients With Gaucher Disease Using Fibroscan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Gaucher_Fibroscan_CTIL
Record Dates: First submitted 2013-03-11; First posted 2013-07-12 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Fibrosis
Keywords: Fibrosis; Gaucher disease
MeSH Terms: conditions — Fibrosis; Gaucher Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Naïve GD patients (Other): Naïve GD patients
  Intervention: device - Fibroscan
  Interventions: Device: Fibroscan
- GD treated with ERT (Other): GD treated with ERT Intervention: device - Fibroscan
  Interventions: Device: Fibroscan
- Healthy control (Other): Healthy control Intervention: device - Fibroscan
  Interventions: Device: Fibroscan
- NonAlcoholic Steatohepatitis Patients (Other): Patients with NonAlcoholic Steatohepatitis( NASH) Intervention: device - Fibroscan
  Interventions: Device: Fibroscan

INTERVENTIONS:
Device: Fibroscan — Fibroscan

SUMMARY:
The investigated cohort will examine liver and spleen fibrosis in patients with Gaucher disease divided into two groups, naive GD patients and GD patients treated with ERT. As liver biopsy in these patients not recommended because the risk of bleeding using Fibroscan is a safe with diagnostic accuracy regarding the liver (& Spleen) fibrosis. Estimating spleen fibrosis is an innovative approach in liver disease and Gaucher.

The evaluation of fibrosis with this new and safe method could avoid complications antiinvasive procedure in GD patients. The addition of fibrosis biomarkers will help for patients score evaluation. The finding of liver and spleen stiffness will be evaluated in native and ERT treated Gaucher patients in order to assess ERT effect on fibrosis.

The Aims are: 1) To assess liver and spleen stiffness measurement using fibroscan and evaluate liver and spleen fibrosis in patients with GD.

2) To compare the elastography in two cohorts of GD patients: ERT treated and naïve GD patients and two control groups of patients: healthy and Non Alcoholic Steatohepatitis (NASH) patients.

3) To correlate the elastography findings with clinical and laboratory data in the four patient groups focusing on Gaucher disease manifestations and GD severity. To compare the elastography in GD naïve and ERT treated patients.

DETAILED DESCRIPTION:
The investigated cohort will include 4 groups of patients 20 probands in each group including: 1) Naïve GD patients 2) GD treated with ERT 3) Healthy control 4) Patients with NonAlcoholic Steatohepatitis( NASH) which are followed at hepatology unit of the Ziv Hospital and healthy controls.

Serum fibrosis markers will be tested including: Bilirubin ,GGT, Haptoglobin,AST,ALT .The findings of spleen and liver fibrosis will be correlated with disease severity usingZimran's Severity Score Index (SSI) liver function tests , serology for viral hepatitis, GDbiomarkers, hemoglobin, platelet levels, and a GD severity score.

Protein C will be measured in all groups of patients Protein C activity as it may be used as a sensitive marker of hepatocellular damage even in those patients with mild liver affection .Also Patients with cirrhosis possess an imbalance in pro-coagulant versus anticoagulantactivity due to increased factor VIII and decreased protein C.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Gaucher in treatment and without treatment.
* Healthy control.
* Patients with Non Alcoholic Steatohepatitis( NASH) which are followed at hepatology unit.

Exclusion Criteria:

• Active liver disease ,cirrhosis patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Liver and spleen fibrosis | 2 years
  Fibrosis will be estimated by the degree of elastography measured by the liver and spleen stifness in kilopascals (kPa).
  Transient elastography will be performed using a Fibro Scan device (EchoSens, Paris, France). A median value [expressed in kilopascals (kPa)] of 10 successful acquisitions will be s considered the representative measurement of liver stiffness. We consider 10 acquisitions with a success rate of at least 60% and an interquartile range (IQR) lower than 20% as representative measurements.
  The FibroScan® and its dedicated probes make up an active, non-implantable medical device using ultrasound. Designed to rapidly measure liver stiffness in a painless and totally non-invasive manner.
  The FibroScan® is based on the one-dimensional pulse elastography technique.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Rosenbaum, Principal Investigator — Rambam Health Corporation